CLINICAL TRIAL: NCT04720664
Title: OASIS: Phase II Trial of OrAl SM-88 in Patients With Metastatic Hormone Receptor-posItive HER2-negative (HR+/HER2-) breaSt Cancer
Brief Title: Oral SM-88 in Patients With Metastatic HR+/HER2- Breast Cancer
Acronym: OASIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Georgetown University (Other)
Collaborators: Tyme, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003282
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Hormone Receptor Positive Breast Carcinoma
Keywords: metastatic; hormone receptor-positive; HER2-negative; breast cancer; oral
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — racemetyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- oral SM-88 (Experimental): SM-88 taken with three conditioning agents: methoxsalen, phenytoin, and sirolimus
  Interventions: Drug: SM-88

INTERVENTIONS:
Drug: SM-88 — * SM-88, Two 230 mg capsules taken orally twice daily (920 mg daily).
  * Methoxsalen, One 10 mg capsule taken orally once daily.
  * Phenytoin, One 50 mg tablet taken orally once daily.
  * Sirolimus, One 0.5 mg tablet taken orally once daily.

SUMMARY:
This is a phase II single arm, open-label study of SM-88 used with methoxsalen, phenytoin, and sirolimus (MPS) in metastatic HR+/HER2- breast cancer. It is designed to determine efficacy, defined as the objective response rate (ORR) of this investigational treatment. It is hypothesized that SM-88 used with MPS will lead to significant anti-tumor responses with acceptable toxicities in patients with metastatic HR+/HER2- breast cancer.

DETAILED DESCRIPTION:
This is a multicenter phase II single arm trial designed to evaluate the efficacy of SM-88 plus three subtherapeutic conditioning agents (methoxsalen, phenytoin, and sirolimus [MPS]) in patients with metastatic HR+/HER2- breast cancer. .

Thirty patients will be enrolled in first stage of the study, and if 3 or more patients have an objective response (complete or partial response) then an additional 20 patients will be enrolled in the second stage of the study. Patients will receive the recommended phase 2 dose (RP2D) of SM-88 (460 mg by mouth [PO] twice a day [BID] D1 - 28) as well as three conditioning agents (MPS): methoxsalen (10 mg PO daily [Qd] D1 - 28), phenytoin (50 mg PO Qd D1 - 28), and sirolimus (0.5 mg PO Qd D1 - 28).

Assessment of efficacy will be conducted every 3 cycles (approximately every 12 weeks) with CT chest/abdomen/pelvis using RECIST v1.1 criteria. Safety including clinic visits, and exams will occur every 4 weeks on Day 1 of each cycle. Laboratory testing will be performed every 2 weeks for the first 2 cycles and then on Day 1 of each subsequent cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer with evidence of metastatic or locally advanced disease, not amenable to resection or radiation therapy with curative intent.
* Documentation of ER-positive and/or PR-positive tumor (≥1% positive stained cells) based on most recent tumor biopsy (discuss with the Principle Investigator if results in different biopsies are discordant in terms of hormone receptor positivity) utilizing an assay consistent with local standards.
* Documented HER2-negative tumor based on local testing on most recent tumor biopsy: HER2-negative tumor is determined as immunohistochemistry score 0/1+ or negative by in situ hybridization (FISH/CISH/SISH) defined by current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines. Patients with equivocal HER2 in situ hybridization results according to current ASCO/CAP guidelines are eligible, as long as they have not received and are not scheduled to receive anti-HER2 treatment.
* Must have progressed on at least 2 lines of endocrine therapy in either the adjuvant or metastatic setting and progressed on a CDK4/6 inhibitor.
* Must have received no more than 4 lines of systemic therapy (for example, including but not limited to endocrine therapy, targeted therapy, biologic therapy, chemotherapy, or experimental therapy) for the treatment of breast cancer in the metastatic setting.
* Premenopausal or postmenopausal female or male patients 18 years of age or older.
* Measurable disease as defined by RECIST v1.1 criteria (tumor ≥ 1 cm in longest diameter on axial image on computed tomography (CT) or magnetic resonance imaging (MRI) and/or lymph node(s) ≥ 1.5 cm in short axis on CT or MRI) on baseline imaging. Bone only metastases must have associated > 10 mm soft tissue mass.
* Asymptomatic brain metastases are allowed if the lesions are not considered to need local therapy. Previously treated brain metastases are allowed as long as they are > 4 weeks from local therapy, clinically asymptomatic, and not requiring high-dose corticosteroids. Patients may remain on steroids for CNS disease if they are taking a stable dose that is less than 10mg of prednisone per day, or the equivalent.
* Must be capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the IRB, prior to the initiation of any screening or study-specific procedures.
* Life expectancy of more than 3 months.
* ECOG performance status 0-1
* Pregnancy must be ruled out in women of childbearing potential. Serum or urine pregnancy test must be negative within 14 days of treatment start in women of childbearing potential and must be willing to have pregnancy test approximately every 4 weeks. Pregnancy testing does not need to be pursued in patients who are judged to be postmenopausal before enrollment, or who have undergone bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation. Patients may be considered postmenopausal in the case that one of the following criteria applies,

  * Prior bilateral oophorectomy, OR
  * Age ≥ 60 years, OR
  * Age < 60 years with intact uterus and amenorrhoeic for ≥ 12 consecutive months prior to chemotherapy and/or endocrine therapy exposure
* Willingness to utilize adequate contraception if of childbearing potential. Women of childbearing potential must use adequate contraception for the duration of protocol treatment and for at least 6 months after the last treatment with SM-88 used with MPS. Adequate contraception is defined as one highly effective form (i.e., abstinence, (fe)male sterilization) OR two effective forms (IUD [non-hormonal preferred], condom with spermicidal foam / gel / film / cream / suppository, occlusive cap with spermicidal foam / gel / film / cream / suppository).
* Must be able and willing to swallow pills whole and retain oral medication.
* Adequate hematologic parameters (Patients must be able to meet the following criteria without transfusion or receipt of colony stimulating factors within 2 weeks before obtaining sample):

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3; Patients must be able to meet the criteria without receipt of colony stimulating factors within 2 weeks before obtaining sample
  * Platelets ≥ 100,000/mm3; Patients must be able to meet the criteria without receipt of transfusion within 2 weeks before obtaining sample
  * Hemoglobin ≥ 9 g/dL; Patients must be able to meet the criteria without receipt of transfusion within 2 weeks before obtaining sample
* Serum creatinine clearance ≥ 60 mL/min based on Cockcroft-Gault equation
* Adequate hepatic parameters:

  * Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) ≤ 3 x ULN (upper limit of normal)
  * Total serum bilirubin ≤ 1.5 x ULN, except for patients with a documented history of Gilbert's Syndrome who can be enrolled at PI discretion
  * For patients with liver metastases, AST and ALT < 5x the institution's ULN and/or total bilirubin ≤ 3.0x the institution's ULN are acceptable as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, or rash.
* Alkaline phosphatase ≤2.5 x ULN (≤5.0 x ULN if bone metastases present)
* Resolution of all acute toxic effects of prior therapy, including radiotherapy to grade ≤1 (except toxicities not considered a safety risk for the patient) and recovery from surgical procedures.
* Must have discontinued all previous therapies for cancer (including endocrine therapy, CDK4/6 inhibitor therapy, cytotoxic chemotherapy, targeted therapy [including, but not limited to, everolimus], radiotherapy, immunotherapy, and investigational therapy) for at least 14 days prior to receiving study drugs and recovered from the acute effects of therapy (treatment-related toxicity resolved to baseline) except for residual alopecia or peripheral neuropathy.

Exclusion Criteria:

* Concurrent therapy with other approved or investigational cancer treatment agents, except bisphosphonates and RANKL inhibitors.
* Bone-only metastases without soft tissue masses measuring > 10 mm.
* Inability to comply with study requirements.
* Diagnosis of other invasive cancer except for adequately treated cervix cancer, or more than 5 years since other diagnosis of invasive cancer (including invasive squamous cell cancers due to contraindication for methoxsalen use) without current evidence of disease.
* Pregnant women or women of childbearing potential without a negative pregnancy test (serum or urine) within 14 days prior to starting study treatment.
* Breastfeeding must be discontinued prior to study entry.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea/vomiting, chronic diarrhea, malabsorption syndrome, intestinal obstruction, or small bowel resection)
* Patients with clinically significant liver disease, including active viral (including hepatitis B, hepatitis C, etc) or other known active hepatitis, current alcohol abuse, or cirrhosis.
* Known chronic hepatitis B virus infection (testing not required prior to enrollment).

  a. Patients with chronic hepatitis C virus infection may be enrolled if there is no clinical/laboratory evidence of cirrhosis per investigator AND the patient's liver function tests fall within the parameters set in the inclusion criteria.
* Uncontrolled HIV infection defined as any of the following 3 criteria: CD4 counts ≤ 350 cells/μL; serum HIV viral load ≥ 400 copies/mL; on a antiretroviral regimen for < 4 weeks prior to treatment with study drugs if anti-retroviral therapy is deemed necessary or appropriate by the investigator.
* Previous enrollment in this study or any other study investigating SM-88.
* History of any known drug allergies to any study medication.
* Clinically significant and uncontrolled major medical condition(s) including, but not limited to uncontrolled nausea/vomiting/diarrhea; active, uncontrolled infection; symptomatic congestive heart failure (New York Heart Association [NYHA] class ≥ II); unstable angina pectoris; cardiac arrhythmia requiring hospitalization in the past 3 months; stroke or MI in the past 6 months.
* Psychiatric illness or social situation that would limit compliance with study requirements.
* Active uncontrolled or symptomatic brain metastases. Previously treated and clinically stable brain metastases, as per Investigator's judgement, are permitted.
* Patients with a seizure disorder that is not well controlled or who have required a change in seizure medications within 60 days of enrollment to the trial.
* Patients with a history of hypersensitivity to phenytoin, its inactive ingredients, or other hydantoins; or a history of prior acute hepatotoxicity attributable to phenytoin.
* Patients treated, or anticipated to be treated, with delavirdine (due to potential for loss of virologic response and possible resistance to delavirdine or to the class of non-nucleoside reverse transcriptase inhibitors caused by phenytoin).
* Patients exhibiting idiosyncratic reactions to psoralen compounds.
* Patients with a history of the light sensitive diseases for which methoxsalen would be contraindicated. Diseases associated with photosensitivity include lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum, and albinism.
* Patients with cutaneous melanoma or invasive squamous cell carcinomas or a history thereof, except for those with stage 1A melanoma or in complete remission for ≥5 years (due to contraindication for use of methoxsalen).
* Patients with a hypersensitivity to sirolimus. Sirolimus does cause immune suppression at the prescribed doses and physicians should note the drugs black box warning to exclude any patient they believe the other exclusion criteria does not reflect.
* Patients with prior allogenic bone marrow transplant or solid organ transplant organ transplant or being treated, or anticipated to be treated, with cyclosporine (because long-term administration of the combination of cyclosporine and sirolimus is associated with deterioration of renal function).
* Patients treated, or anticipated to be treated, with a calcineurin inhibitor (because concomitant use of sirolimus and a calcineurin inhibitor increases the risk of calcineurin inhibitor-induced hemolytic uremic syndrome/thrombotic thrombocytopenic purpura/thrombotic microangiopathy [HUS/TTP/TMA]).
* Current use of known strong inhibitors or inducers of CYP3A4, CYP2C9 or CYP2C19 within 14 days of initiation of study drug. When possible these medications and grapefruit juice should be avoided for the duration of the study treatment and alternate therapies are preferred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ashai, MD, Principal Investigator — Georgetown University
Locations (5):
- United States (5):
  - MedStar Georgetown University Hospital, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral SM-88: SM-88 taken with three conditioning agents: methoxsalen, phenytoin, and sirolimus
  SM-88: • SM-88, Two 230 mg capsules taken orally twice daily (920 mg daily).
  * Methoxsalen, One 10 mg capsule taken orally once daily.
  * Phenytoin, One 50 mg tablet taken orally once daily.
  * Sirolimus, One 0.5 mg tablet taken orally once daily.
Period: Overall Study
Arm/Group | Oral SM-88
Started | 11
Completed | 0
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 9

BASELINE CHARACTERISTICS:
Arm/Group | Oral SM-88
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Anti-tumor efficacy will be defined as partial response (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 for target lesions assessed by CT or MRI. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 8 weeks until progression (an average of 8 weeks)
Population: No patients responded to treatment on the first assessment.
Measure: Number; unit: percentage of patients
Arm/Group | Oral SM-88
Number analyzed (Participants) | 11
percentage of patients | 0

2. Secondary Outcome: Duration of Response (DOR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 for target lesions assessed by CT or MRI. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 8 weeks until Progression (an average of 8 weeks)
Population: Outcome unable to be analyzed since there were no participants with a response.
Arm/Group | Oral SM-88
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time in days from study entry to the first documented disease progression per RECIST v1.1 as assessed by local site or death. Patients who are alive and free from progression on the date of closing follow-up will be censored on that date.
Time Frame: Every 8 weeks until progression (an average of 8 weeks)
Population: Median measure is in days.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oral SM-88
Number analyzed (Participants) | 11
days | 51 [28 to 79]

4. Secondary Outcome: Clinical Benefit Rate (CBR) at ≥ 24 Weeks
Description: The percentage of patients who have complete response (CR), partial response (PR), or stable disease (SD) at ≥ 24 weeks will be reported.
Time Frame: 24 weeks
Population: No participants were on trial at 24 weeks so outcome can not be analyzed.
Arm/Group | Oral SM-88
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Treatment-Related Adverse Events [Safety and Tolerability]
Description: The number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Time Frame: From the time of the administration of study drug until discontinuation of therapy (every 4 weeks on Day 1 of each cycle in a 28 day cycle; approximately 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral SM-88
Number analyzed (Participants) | 11
Participants | 6

ADVERSE EVENTS:
Time Frame: From the time of the administration of study drug until discontinuation of therapy (every 4 weeks on Day 1 of each cycle in a 28 day cycle; approximately 3 months)
Arm/Group | Oral SM-88
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral SM-88 (N=11)
Infections and infestations - Other, specify (Investigations) | 1 (1) — Increased Liver Function Tests
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral SM-88 (N=11)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (7)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Weakness
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — COVID infection
Upper respiratory infection (Infections and infestations) | 1 (1) — COVID +
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 7 (11)
Blood bilirubin increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Skin and subcutaneous other- discoloration of lower extremities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT04720664/Prot_SAP_000.pdf